CLINICAL TRIAL: NCT06603714
Title: Immediate Effects of Instrument Assisted Soft Tissue Mobilization at Different Muscle Lengths
Brief Title: Effects of Soft Tissue Mobilization at Different Muscle Lengths
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, Matej Voglar, Assistant professor, University of Primorska
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IASTM_effects
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Muscle, Ligament and Fascia Disorders; Instrument Assisted Soft Tissue Mobilization; Range of Motion; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Each participant will complete two visits. During one visit the treatment will be performed at short, whilst during the other at long muscle lengths.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated segment - stretched (Experimental): Instrument assisted soft tissue mobilization will be completed with the calf muscles in a shortened position (30° knee flexion and full ankle plantar flexion).
  Interventions: Other: Instrument assisted soft tissue mobilization
- Treated segment - shortened (Experimental): Instrument assisted soft tissue mobilization will be completed with the calf muscles in a lengthened position (full knee extension and approximately 0° ankle dorsiflexion).
  Interventions: Other: Instrument assisted soft tissue mobilization

INTERVENTIONS:
Other: Instrument assisted soft tissue mobilization — We will perform instrument assisted soft tissue mobilization on calf muscles. The intervention will last 9 min. For the first minute of treatment light pressure will be applied for tissue preparation. Afterwards, four different strokes will be applied by maintaining the tool at a 30° of inclination for one minute. This will be repeated for a second set, with a tool inclination of 45°.
  Other Names: Stretching

SUMMARY:
The purpose of this study will be to compare the effects of instrument assisted soft tissue mobilization at different muscle lengths on pain pressure thresholds and measures of flexibility.

DETAILED DESCRIPTION:
Instrument assisted soft tissue mobilization is a widely used manual therapy technique, which aims at reducing pain and improving range of motion. Evidence regarding acute responses to instrument assisted soft tissue mobilization at different muscle lengths is lacking. Therefore, the purpose of our study was to conduct a cross-over trial and compare the acute effects of instrument assisted soft tissue mobilization at short and long muscle lengths of the calf muscles on pain pressure thresholds and measures of flexibility.

ELIGIBILITY:
Inclusion Criteria:

* without previous lower limb injuries in the last year
* healthy individuals
* students

Exclusion Criteria:

* Patients with acute lower limb disorders e.g. open wounds, hematoma, trauma
* General hypermobility: Beighton score >4.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-05 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Pain pressure threshold | 30 minutes
  Pain pressure threshold will be measured via handheld algometer on the proximal third of the distance between medial condyle of the femur and lateral malleolus.
Passive dorsiflexion range of motion | 30 minutes
  Passive dorsiflexion will be measured via two wooden boards connected with a hinge. We will apply a standardized torque of 30,9 Nm via handheld dynamometer. Each visit, participants will be measured before and after the performed intervention.

SECONDARY OUTCOMES:
Stand and reach test | 30 minutes
  With the help of a standardized measuring tool, participants will activelly bend as low as possible.
Lumbar spine flexibility | 30 minutes
  Sagittal profile of the spine will be measured measured via device: Idiag M360 (MediMouse, Idiag AG, Fehraltorf, Switzerland). End range of motion of the whole lumbar spine was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Primorska, Faculty of Health Sciences, Izola, Primorska, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided